CLINICAL TRIAL: NCT01308320
Title: Dose-dependent Effect of Fentanyl on Cough Attenuation During Emergence From General Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jeong-Rim Lee / Assistant Professor, Severance Hospital, Department of Anesthesiology and Pain Medicine in Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2009-0111
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Thyroid Neoplasm
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- saline (Placebo Comparator): control group
  Interventions: Drug: saline
- F1 group (Active Comparator): F1 group : fentanyl 1 mcg/kg
  Interventions: Drug: fentanyl citrate
- F1.5 group (Active Comparator): F1.5 group : fentanyl 1.5 mcg/kg
  Interventions: Drug: fentanyl citrate
- F2 group (Active Comparator): F2 group : fentanyl 2 mcg/kg
  Interventions: Drug: fentanyl citrate

INTERVENTIONS:
Drug: fentanyl citrate — According to the enrolled group, certain dose of fentanyl is intravenously administered by bolus just after sevoflurane discontinuation.
  Arms: F1 group; F1.5 group; F2 group
Drug: saline — According to the enrolled group, certain dose of saline is intravenously administered by bolus just after sevoflurane discontinuation.
  Arms: saline

SUMMARY:
Fentanyl is expected to suppress tracheal tube-induced cough during emergence from general anaesthesia through binding to its receptors in the brainstem. However, it has not been proven if fentanyl has a complication-free, dose-dependent effect on cough suppression during emergence from sevoflurane anaesthesia. The purpose of this study is to evaluate the relationship between fentanyl doses and cough suppression during emergence from sevoflurane anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* the patients undergoing general anaesthesia for elective thyroidectomy due to thyroid neoplasm.
* ASA I-II.
* 20-59 years old.
* female only.

Exclusion Criteria:

* signs of difficult intubation.
* risks for perioperative pulmonary aspiration.
* history of chronic respiratory disease.
* recent upper respiratory track infection.
* previous and recent smoking history

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Tagaito Y, Isono S, Nishino T. Upper airway reflexes during a combination of propofol and fentanyl anesthesia. Anesthesiology. 1998 Jun;88(6):1459-66. doi: 10.1097/00000542-199806000-00007. PMID 9637637
- [Background] Nishina K, Mikawa K, Maekawa N, Obara H. Fentanyl attenuates cardiovascular responses to tracheal extubation. Acta Anaesthesiol Scand. 1995 Jan;39(1):85-9. doi: 10.1111/j.1399-6576.1995.tb05597.x. PMID 7725888